CLINICAL TRIAL: NCT06666218
Title: Helping Ovarian Cancer Patients Cope With Their Disease (HOPE) - Phase 2
Brief Title: Helping Ovarian Cancer Patients Cope With Their Illness (HOPE)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment is currently paused. Aim 1 recruitment has finished, and the study team is preparing to begin Aim 2 recruitment.
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1124787; NCI-2024-08640 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20682 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Behavior Therapy; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aim 1 (HOPE intervention workshop, survey, interview) (Experimental): Patients complete the HOPE intervention workshop virtually or in person. The workshop consists of three weekly sessions, each lasting 60 to 90 minutes, along with a survey and an interview for HOPE Intervention refinement during follow up.
  Interventions: Behavioral: Behavioral Intervention; Other: Electronic Health Record Review; Other: Interview; Other: Survey Administration
- Aim 2, Group I (HOPE intervention workshop) (Experimental): Patients complete the HOPE intervention workshop either virtually or in person, with three weekly sessions, each lasting 60 to 90 minutes.
  Interventions: Behavioral: Behavioral Intervention; Other: Electronic Health Record Review; Other: Survey Administration
- Aim 2, Group II (usual care) (Active Comparator): Patients receive usual care on study.
  Interventions: Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Complete the HOPE intervention workshop
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Lifestyle Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Aim 1 (HOPE intervention workshop, survey, interview); Aim 2, Group I (HOPE intervention workshop)
Other: Electronic Health Record Review — Ancillary studies
Other: Interview — Complete an interview
  Arms: Aim 1 (HOPE intervention workshop, survey, interview)
Other: Survey Administration — Complete a survey
  Arms: Aim 1 (HOPE intervention workshop, survey, interview)
Other: Survey Administration — Ancillary studies
  Arms: Aim 2, Group I (HOPE intervention workshop); Aim 2, Group II (usual care)

SUMMARY:
This clinical trial compares the effect of the Helping Ovarian Cancer Patients Cope with Their Disease (HOPE) intervention to usual care for the reduction of hopelessness and helplessness in patients with ovarian cancer that has come back after a period of improvement (recurrent). Patients with recurrent ovarian cancer are at high risk for increased death and poor mental health outcomes, including depression and anxiety. Ovarian cancer is the deadliest of all gynecologic cancers, with a survival rate at five years of only 50%. Most patients are diagnosed with advanced disease and have a high chance of recurrent disease that is incurable, even if upfront treatments are effective. Ovarian cancer's advanced diagnosis, high likelihood of recurrence and death, and rigorous treatment including surgery and other cancer therapies create high levels of distress and reduced quality of life (QOL). Patients with recurrent ovarian cancer report high rates of depression and anxiety and poor QOL. Due to the major distress, reduced QOL, and likelihood of death among this population, improving this patient population's QOL is a priority. Using the HOPE intervention may be effective in reducing hopelessness and helplessness in recurrent ovarian cancer patients.

DETAILED DESCRIPTION:
OUTLINE:

AIM 1: Patients complete the HOPE intervention workshop virtually or in-person. The workshop consists of 3 sessions, each held once per week and lasting 60 to 90 minutes as well as complete a survey and an interview for HOPE intervention refinement during follow up.

AIM 2: Patients are randomized to 1 of 2 groups.

GROUP I: Patients complete the HOPE intervention workshop virtually or in-person, with 3 sessions held once per week, each lasting 60 to 90 minutes.

GROUP II: Patients receive usual care on study.

Patients in both groups complete baselines and follow up assessments 5, 8, and 12 weeks after the randomization event.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* English speaking
* Able to provide informed consent
* Current diagnosis of recurrent epithelial ovarian cancer (regardless of the amount of time since the diagnosis, given the poor prognosis of this illness with a median survival time of less than 2 years)

Exclusion Criteria:

* Patients with non-invasive gynecologic disease (i.e., dysplasia)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Accrual rates (Aim 1) | At the time of enrollment
  Feasibility will be assessed by accrual rates. Feasibility cutoffs will include >= 50% of eligible patients will enroll in the study.
Fidelity rates (Aim 1) | Up to 28 days
  Feasibility will be assessed by fidelity rates. Feasibility cutoffs will include >= 75% of HOPE workshop sessions delivered with fidelity.
Rates of intervention completion (Aim 1) | Up to 28 days
  Feasibility will be assessed by rates of intervention completion (all three sessions of Helping Ovarian Cancer Patients Cope with Their Disease [HOPE]). Feasibility cutoffs will include 70% of enrolled patients will complete all workshop sessions.
Acceptability of the HOPE intervention (Aim 1) | Up to 28 days
  Acceptability will be assessed by the Theoretical Framework of Acceptability (TFA) questionnaire, which is an 8-item questionnaire assessing acceptability of healthcare interventions across seven constructions: affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness and self-efficacy. The eighth item is a general acceptability item. Items are rated on a 5-point Likert scale (e.g., 1 = strongly dislike, 5 = strongly like) and a mean is computed across all seven constructs and a single outcome is examined for the general item. Scores on the TFA questionnaire will be calculated using the total mean score of seven TFA items. A single-item score will be used for the remaining eighth item, which is a general item assessing acceptability. In this study, will use a cutoff of >= 70% agreeing (or rating as confident, liking, acceptable) as being acceptable for use.
Overall satisfaction (Aim 1) | Up to 28 days
  Satisfaction will be assessed by using three items assessing overall satisfaction (How satisfied are you? How likely are you to recommend to someone? How likely would you participate in this workshop knowing what it is like now?). A cutoff score of >= 7 (out of 10) will be used as a cutoff for each satisfaction item.
Change in hopelessness/helplessness (Aim 2) | Baseline to 12 weeks post-randomization
  Hopelessness/helplessness will be measured by the helplessness/hopelessness subscale of the Mental Adjustment to Cancer (MAC) scale. The MAC scale is a widely used, 40-item scale that assesses patients' psychological responses to cancer. Items are given as statements (e.g., "I feel that life is hopeless") and patients report their agreement using a 4-point Likert-scale (1 = definitely does not apply to me, 2 = does not apply to me, 3 = applies to me, 4 = definitely applies to me).

SECONDARY OUTCOMES:
Accrual rates (Aim 2) | At the time of enrollment
  Feasibility will be assessed by accrual rates. Feasibility will be examined by conducting frequency and descriptive statistics for enrollment rates. The benchmark for feasibility is >= 50% of screened eligible patients enroll in the study. Feasibility process outcomes will be analyzed to determine whether the intervention is feasible for future dissemination and implementation efforts and recruitment of a full-scale randomized controlled trial (RCT) as well as to determine engagement.
Rates of intervention completion (Aim 2) | Up to 35 days
  Feasibility will be assessed by rates of intervention completion (all three sessions of HOPE). Feasibility will be examined by conducting frequency and descriptive statistics for intervention workshop completion. The benchmark for feasibility is >= 70% of enrolled patients will complete the intervention (e.g., complete all workshop sessions). Feasibility process outcomes will be analyzed to determine whether the intervention is feasible for future dissemination and implementation efforts and recruitment of a full-scale RCT as well as to determine engagement.
Acceptability of the HOPE intervention (Aim 2) | 5-weeks post-randomization
  Acceptability will be assessed by the TFA questionnaire, which is an 8-item questionnaire assessing acceptability of healthcare interventions across seven constructions: affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness and self-efficacy. The eighth item is a general acceptability item. Items are rated on a 5-point Likert scale (e.g., 1 = strongly dislike, 5 = strongly like) and a mean is computed across all seven constructs and a single outcome is examined for the general item. A cutoff of 70% will be used to assess acceptability. If < 70% agree/rate as acceptable, this indicates modification of the protocol. If >= 70% agree/rate as acceptable, this indicates no modification of the protocol.
Change in distress (Aim 2) | Baseline to 5 weeks post-randomization
  Distress will be assessed using two measures. (1) The Patient Health Questionnaire which is an 8-item questionnaire assessing depression on a 4-point Likert scale (0 = not at all, 3 = nearly every day). (2) The Generalized Anxiety Disorder, which is a 7-item self-report anxiety measure asking about how commonly feelings of anxiety are experienced (0 = not at all, 3 = nearly every day), will be used to assess anxiety.
Change in quality of life (QOL) (Aim 2) | Baseline to 5 weeks post-randomization
  QOL will be assessed using the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) scale. The FACT-O is a 39-item, validated scale that assesses the five domains of QOL among ovarian cancer patients: physical, functional, social/family, emotional, and additional concerns related to ovarian cancer. All items are rated on a 5-point Likert scale (0 to 4), with higher scores indicating higher levels of QOL. Will use mixed effects models (linear and logistic). The mixed models will have a patient-level random intercept, fixed effects for time trend parameter(s), treatment and treatment x time interaction. All analyses will be intention-to-treat. Will set α=0.05 and adjust type I error using Holm's stepdown procedure.
Change in self-efficacy for treatment decision-making (Aim 2) | Baseline to 5 weeks post-randomization
  Self-efficacy for treatment decision-making will be measured by Decision-Making Participation Self-Efficacy (DEPS) scale. The DEPS scale is a 5-item validated measure that assesses cancer patients' confidence in engaging in difference activities related to decision-making. Patients are asked to indicate how confident they are that they would be able to engage in various decision-making activities (e.g., "Tell your doctor about the option you would prefer"); items are rated on a 5-point Likert scale (1 = not at all confident, 5 = completely confident). Will use mixed effects models (linear and logistic). The mixed models will have a patient-level random intercept, fixed effects for time trend parameter(s), treatment and treatment x time interaction. All analyses will be intention-to-treat. Will set α=0.05 and adjust type I error using Holm's stepdown procedure.
Change in readiness for advance care planning (ACP) (Aim 2) | Baseline to 5 weeks post-randomization
  Engagement in ACP will be measured by readiness for ACP using the reliable and valid Advance Care Planning Readiness Scale to assess readiness for end-of-life care conversations. This is an 8-item measure, which is scored on a Likert scale (1 = strongly disagree, 7 = strongly agree), with higher scores indicating increased overall readiness to engage in ACP by discussing and making end-of-life care decisions.
Change in level of engagement in advance care planning (ACP) (Aim 2) | Baseline to 5 weeks post-randomization
  Engagement in ACP will be measured by level of engagement in ACP using the reliable and valid Advance Care Planning Engagement Survey: Action Measures. This scale is composed of four sub-scales with a total of 18 items. All items are rated on a yes=1 and no=0. Scores can range from 0 (no action taken) to 18 (all actions taken). Higher scores indicate greater engagement in ACP.
Change in documentation of advance care planning (ACP) conversations (Aim 2) | Baseline to 5 weeks post-randomization
  Engagement in ACP will be measured by documentation of ACP conversations using an 8-item measure of discussing end-of-life care, living will, health care proxy (HCP), and do-not-resuscitate (DNR) orders with family and doctor. All items are yes/no questions (yes = 1, no = 0). Items are summed to provide an overall measure of ACP conversations from 0 (no conversations) to 8 (all conversations with family and doctors).
Change in completion of advance care directives (Aim 2) | Baseline to 5 weeks post-randomization
  This will be assessed by asking patients whether they have completed a Do Not Resuscitate (DNR) order, living will, or identified a health care proxy (HCP). All items are yes/no questions (yes = 1, no =0). Items are summed to provide an overall measure of 0 (no advance directives) to 3 (all advance directives completed).

CONTACTS AND LOCATIONS:
Overall Officials: Megan J. Shen, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No